CLINICAL TRIAL: NCT02392728
Title: The Effectiveness of Virtual Environment on the Adverse Psychological Effects in Patients Receiving Treatment for Cancer
Brief Title: Virtual Environments in Patients Receiving Treatment for Cancer
Acronym: VE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Collaborators: University of Cyprus (Other)
Responsible Party: Principal Investigator, Dr. Andreas Charalambous, Assistant Professor, Cyprus University of Technology
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AC-VES-91
Record Dates: First submitted 2015-03-06; First posted 2015-03-19 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Mood Disturbances
MeSH Terms: interventions — Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention VE (Experimental): Session of Immersive Virtual Reality (VR) and Session of Guided Imagery
  Interventions: Behavioral: Immersive Virtual Reality (VR); Behavioral: Guided Imagery
- Intervention GI (Active Comparator): Session of Immersive Virtual Reality (VR) and Session of Guided Imagery
  Interventions: Behavioral: Immersive Virtual Reality (VR); Behavioral: Guided Imagery

INTERVENTIONS:
Behavioral: Immersive Virtual Reality (VR) — Patients in this group will experience the virtual content (e.g., natural scenes) through a Head-Mounted-Display, simulating movement by manipulating a gesture controller. Following a resting period the patients will then experience the guided imagery session (e.g. visual images of pleasant scenery)
Behavioral: Guided Imagery — Patients in this group will experience the guided imagery (e.g. visual images of pleasant scenery). Following a resting period the patients will then experience the virtual content (e.g., natural scenes) through a Head-Mounted-Display, simulating movement by manipulating a gesture controller

SUMMARY:
The mood disturbances that lung cancer patients experience during and after chemotherapy have a debilitating effect on their quality of life. The goal of the proposed project is to develop and test an intervention that relies on the use of immersive Virtual Reality (VR) to combat the adverse psychological/emotional consequences of receiving treatment for cancer. Although VR has been used with success to treat various psychological conditions (e.g., phobias, PTSD), its potential in helping cancer patients experience an improved mood and hence better quality of life has not yet been tested. In this project the investigators will first develop the virtual content (e.g., natural scenes) that patients will experience within a Head-Mounted-Display, simulating movement by manipulating a gesture controller. The investigators will then carry out a randomized, double blind, crossover trial with 50 hospitalized cancer patients to test whether they can benefit psychologically and emotionally from their interaction with an immersive environment compared to those who will experience a guided imagery intervention. A positive result will open the route for the future development of affordable self-administered VR solutions for treating the psychological side-effects of cancer treatment.

DETAILED DESCRIPTION:
Although VR has been used with success to treat various psychological conditions (e.g., phobias, PTSD), its potential in helping cancer patients experience an improved mood and hence better quality of life has not yet been tested. In this project the investigators will first develop the virtual content (e.g., natural scenes) that patients will experience within a Head-Mounted-Display, simulating movement by manipulating a gesture controller. The investigators will then carry out a randomized, double blind, crossover trial with 50 hospitalized cancer patients to test whether they can benefit psychologically and emotionally from their interaction with an immersive environment compared to those who will experience a guided imagery intervention. A positive result will open the route for the future development of affordable self-administered VR solutions for treating the psychological side-effects of cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they had a histopathological diagnosis of cancer (different types are allowed)
* were 18 years or older, on active treatment and were receiving care at the hospital as inpatients
* Eligible participants will need to be able to speak and understand Greek and they had given written informed consent
* Participants should also have a score of >60 on the POMS total mood disturbance scale, a >50 on the Karnofsky Performance Scale Index
* a mean of >50 on the Attentional Function Index (AFI)

Exclusion Criteria:

* Patients were excluded if they were receiving palliative care
* they had an impaired cognitive ability or
* they had an impaired visual ability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Changes in Mood Disturbances as measured by the POMS | Baseline and then participants will be followed for the duration of the intervention, an expected average of 8 days
  The POMS total mood disturbance comprises subscales that evaluate anxiety, depression, anger, vigor, fatigue, and confusion. The possible range of scores for the TMDS is -40 through 192 with higher scores indicating greater mood. Lower scores indicate an improvement in mood

SECONDARY OUTCOMES:
Changes in Quality of Life as measured by FACT-G | Baseline and then participants will be followed for the duration of the intervention, an expected average of 8 days
  FACT-G, is a self-report instrument consisting of 27-items
Changes in Blood Pressure | Baseline and then participants will be followed for the duration of the intervention, an expected average of 8 days
  Measurement of Blood Pressure
Changes in Heart Rate | Baseline and then participants will be followed for the duration of the intervention, an expected average of 8 days
  Measurement of Heart Rate

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Charalambous, Principal Investigator — andreas.charalambous@cut.ac.cy
Locations (1):
- American Medical Centre, Nicosia, Cyprus

REFERENCES:
- [Derived] Ioannou A, Paikousis L, Papastavrou E, Avraamides MN, Astras G, Charalambous A. Effectiveness of Virtual Reality Vs Guided Imagery on mood changes in cancer patients receiving chemotherapy treatment: A crossover trial. Eur J Oncol Nurs. 2022 Dec;61:102188. doi: 10.1016/j.ejon.2022.102188. Epub 2022 Aug 13. PMID 36202024